CLINICAL TRIAL: NCT00866060
Title: Donepezil and Memantine in Moderate to Severe Alzheimer's Disease
Acronym: DOMINO-AD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Dr Gill Dale, King's College London
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006/123; ISRCTN49545035; Eudract 2007-001172-36
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Moderate to Severe Alzheimer's Disease
Keywords: donepezil; memantine; moderately severe Alzheimer's disease; severe Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): 10mg donepezil plus 20mg memantine
  Participants in this arm will continue with their current donepezil 10mg/day regimen and immediately commence active memantine at a dose of 5mg per day, increasing in 5mg increments weekly until 20mg per day is achieved from week 4 onwards
  Interventions: Drug: Memantine; Drug: Donepezil
- 2 (Placebo Comparator): Placebo donepezil plus 20mg memantine
  Participants in this arm will immediately commence active memantine at a dose of 5mg per day, increasing in 5mg increments weekly until 20mg per day is achieved from week 4 onwards. Donepezil dose will be reduced to 5mg daily in weeks 1 to 4 and replaced with placebo donepezil in week 5.
  Interventions: Drug: Memantine; Drug: Placebo donepezil
- 3 (Placebo Comparator): 10mg donepezil plus placebo memantine
  Participants in this arm will continue with their current donepezil 10mg/day regimen and immediately commence placebo memantine.
  Interventions: Drug: Donepezil; Drug: Placebo memantine
- 4 (Placebo Comparator): Placebo donepezil plus placebo memantine
  Participants in this arm will immediately commence placebo memantine dose escalation and will switch to donepezil 5mg daily in weeks 1 to 4, and replaced with placebo donepezil in week 5.
  Interventions: Drug: Placebo donepezil; Drug: Placebo memantine

INTERVENTIONS:
Drug: Memantine — 20mg memantine
  Other Names: Ebixa
  Arms: 1; 2
Drug: Donepezil — 10mg donepezil
  Other Names: Aricept
  Arms: 1; 3
Drug: Placebo donepezil — Placebo donepezil
  Arms: 2; 4
Drug: Placebo memantine — Placebo memantine
  Arms: 3; 4

SUMMARY:
The trial will examine whether pharmacological treatment with donepezil, memantine or combination of memantine and donepezil is any better than a placebo (dummy) treatment in people with Alzheimer's disease who have reached the moderate to severe stage of illness. Using a double blind design, where neither the investigators nor participants know who is receiving which treatment, participants will be randomly assigned to one of these four treatment groups (donepezil and memantine, memantine only, donepezil only or placebo). In order to keep both the investigators and participants blind to drug allocation a double dummy design will be necessary. This means that each participant will receive 2 treatments - either an active form or placebo of each of the 2 study drugs.

Hypotheses are:

1. Patients with Alzheimer's disease (AD) who continue donepezil beyond the point of transition from moderate to severe dementia continue to show significantly less decline on ratings of cognitive function and activities of daily living over the following 12 months than those discontinuing donepezil.
2. Patients with AD who change to memantine therapy in place of donepezil at the point of transition from moderate to severe dementia show significantly smaller decline on ratings of cognitive function and activities of daily living over the following 12 months than those who receive placebo.
3. Patients given the combination of memantine and donepezil at the point of transition from moderate to severe dementia show significant additive or synergistic benefits on measures of activities of daily living and cognitive function after 12 months compared to those patients continuing on either drug as a single treatment.

DETAILED DESCRIPTION:
This trial will involve the withdrawal of drug participants that are currently on (donepezil) and in arm 4, the participant will only be on placebo treatment. It is important to include this arm of the study as a key objective in looking at the benefit of continuing donepezil and therefore a placebo arm should be present as a comparator. To reduce the risk to participants of withdrawing donepezil too early in their illness, an inclusion criteria is that the participant is at a stage in their disease whereby the prescribing clinician feels a change in drug prescription may be appropriate.

ELIGIBILITY:
Inclusion Criteria:

Participants will be patients who meet NINCDS-ADRDA criteria for probable or possible Alzheimer's disease (McKhann et al, 1984). In addition they will meet all of the following criteria:

1. SMMSE = 5 to 13 (13 chosen as NICE threshold of 10 plus 1 SD on SMMSE score)
2. Continuously prescribed donepezil for at least 3 months
3. Maintained on 10mg donepezil in previous 6 weeks.
4. No changes in prescription of any psychotropic (antipsychotic, antidepressant, benzodiazepine) medication in previous 6 weeks.
5. Prescribing clinician considers (based on NICE guidance, discussions with patient and carer and clinical judgement) that change of drug treatment (i.e. stop donepezil or introduce memantine) may be appropriate.
6. Patient is community resident and has family or professional carer or is visited on at least a daily basis by carer.
7. Patient agrees to participate if considered capable (see section 7.5)
8. Main carer (informal or professional) consents to their own involvement and the patient's involvement -

Exclusion Criteria:

To maximise the generalisability of the study data, exclusions will be kept to a minimum. These will include:

1. Patient has severe, unstable or poorly controlled medical conditions apparent from physical examination or clinical history.
2. Patient is already prescribed memantine.
3. Patient is unable to take trial medications because of contra-indications or previous adverse or allergic reactions.
4. Patient is involved in another clinical trial.
5. Clinician considers patient would not be compliant with trial medication. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2008-02; Primary Completion 2012-02 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function measured with the Standardised MMSE (SMMSE). | 4 years
Activities of Daily Living measured with the Bristol Activities of Daily Living scale (BADLS). | 4 years

SECONDARY OUTCOMES:
Non-cognitive dementia symptoms measured with the Neuropsychiatric Inventory (NPI) and the Cohen-Mansfield Agitation Inventory. | 4 years
Health-related quality of life measured with the EQ-5D (Euroqol Group 1990) and the DEMQOL-Proxy (Smith et al 2004) - a carer-rated and disease-specific measure of quality of life in dementia. | 4 years
Care-giver burden measured with the General Health Questionnaire. | 4 years
Cost effectiveness assessed through consideration of the combination of costs generated from the Client Service Receipt Inventory (CSRI) and the assessments of function and quality of life (BADLS, DEMQOL, EQ-5D). | 4 years
Institutionalisation defined as permanent transition from living in an independent household to a care home, NHS continuing care unit or hospital and measured with questions taken from the CSRI and telephone interviews. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Howard, MD, Principal Investigator — Institute of Psychiatry
Locations (1):
- Institute of Psychiatry, London, United Kingdom